CLINICAL TRIAL: NCT06025968
Title: Digital Cognitive-behavioral Therapy for Insomnia for Patients With Multiple Sclerosis: A Randomised Controlled Trial
Brief Title: Digital Cognitive-behavioral Therapy for Insomnia for Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Monica Buhrman, Associate professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uppsala univerisity
Record Dates: First submitted 2023-08-20; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis; Insomnia
MeSH Terms: conditions — Multiple Sclerosis; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be adiministered via a digital platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-CBT (Experimental): Cognitive behavioral therapy for insomnia with adjustment for MS.
  Interventions: Behavioral: i-CBT
- Applied relaxation (Active Comparator): Applied relaxation with adjustments for MS.
  Interventions: Behavioral: Applied relaxation

INTERVENTIONS:
Behavioral: i-CBT — The content is based on manual by Perlis et al (2015) and has slightly reworked by the research team by shortening treatment from seven to six sessions and allowing for day-time naps that may be necessary for patient with MS (Siengsukon et al. 2020). Due to the high prevalence of fatigue in people with MS, naps during the day may be a necessity to cope with everyday tasks. In cases where patients could not refrain from naps, they were advised to limit them to maximum 20 minutes and to take them as early in the day as possible. Other components are sleep restriction, sleep hygiene, stimulus control and cognitive techniques..
  Arms: i-CBT
Behavioral: Applied relaxation — Treatment consits of 6 modules. The main components in the training program will be progressive muscle relaxation, short relaxation with release only and without tension, and finally the participants will be taught rapid relaxation.
  Arms: Applied relaxation

SUMMARY:
The goal of this clinical trialis to compare a digital Cognitive-behavioral intervention for insomnia to digital administered applied relaxation in participants with Multiple Sclerosis.

The treatments will be compared in following outcomes:

* Sleep diary: total sleep time (TST), sleep onset latency (SOL), wake after sleep onset (WASO), and early morning awakening (EMA).
* Insomnia symptoms
* Depressive symptoms
* Client satisfaction
* Negative effects
* Worry
* Fatigue
* Quality of life
* MS symptoms/function

DETAILED DESCRIPTION:
In order to start evaluate the digital treatment format, this study will use a Randomized Controlled Trial design (RCT). Participants with MS and insomnia from a Neurology clinic in Sweden will be randomized to either Cognitive-behavioral intervention for insomnia (iCBT) or Applied relaxation (AR). The treatments will consits of six sessions and will be administered digitally. Psychologists will have contact with the participants via a secure video call platform.Follow-up data will be gathered at six and 12 months after the treatments.

The treatments will be compared in following outcomes:

* Sleep diary: total sleep time (TST), sleep onset latency (SOL), wake after sleep onset (WASO), and early morning awakening (EMA).
* Insomnia symptoms
* Depressive symptoms
* Worry
* Fatigue
* Quality of life
* MS symptoms/function
* Client satisfaction
* Negative effects

ELIGIBILITY:
Inclusion Criteria:

* be medically assessed
* meet criteria for MS and insomnia disorder
* have access to the internet and a smart phone with internet access
* have good reading ability, and
* be over 18 years of age

Exclusion Criteria:

* have a planned treatment that may prevent participation
* were involved in ongoing medical research that may prevent participation,
* do not have a command of the Swedish language
* have a more serious acute psychiatric and/or somatic condition which prevented participation; or benefit from the treatment
* have an increased risk of suicide to the extent that participation in study was considered inappropriate,
* suffers from other primary sleep disorders such as sleep apnea, restless legs syndrome, periodic limb movement disorder, circadian rhythm disorder, or parasomnia
* have insomnia due to environmental factors such as shift work.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Sleep diary - Total Wake Time (TWT) | Baseline, daily through study completion, up to 8 weeks
  Total wake time (TWT) is calculated by summing the variables Sleep onset latensy, Wake after slepp onset and Early morning awakening in minutes from the sleep diary. This measure has been used as an outcome measure in clinical studies of CBT-I because it may have better explanatory power than other variables in the sleep diary. .

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline (before the treatment) after the treatment that is 6 to 8 weeks after entering the treatment, and 6 and 12 months after the treatment.
  Measures the severity of insomnia and consists of seven questions regarding the individual's experience of insomnia with response options on a five-point Likert scale from 0-4. HIgher values indicating more severe insomna.
Patient Health Questionnaire (PHQ-9) | Baseline (before the treatment) after the treatment that is 6 to 8 weeks after entering the treatment and 6 and 12 months after the treatment.s.
  The PHQ-9 consists of nine questions designed according to diagnostic criteria for major depression in the DSM-5, as well as a question on level of functioning.Higher values indicating worse outcome.
The Generalized Anxiety Disorder (GAD-7) | Baseline (before the treatment) after the treatment that is 6 to 8 weeks after entering the treatment and 6 and 12 months after the treatment.
  Questionnaire which is a seven-item, self-report anxiety questionnaire designed to assess feelings of anxiety and worrying (Spitzer 2006). Each item is scored on a Likert scale between 0 and 3 and totaled for a score of 0 to 21. Higher score indicating worse outcome.
Fatigue Severity Scale (FSS) | Baseline (before the treatment) after the treatment that is 6 to 8 weeks after entering the treatment and 6 and 12 months after the treatment.
  Consists of nine questions with response options on a seven-point Likert scale 1 - 7 (Krupp et al, 1989). The total score is divided by the number of questions to give a mean score between 1 - 7. The higher the score, the more severe the fatigue..
The Brunnsviken Brief Quality of Life Scale (BBQ) | Baseline (before the treatment) after the treatment that is 6 to 8 weeks after entering the treatment, and 6 and 12 months after the treatment.
  The BBQ comprise twelve items corresponding to satisfaction and importance of six life areas (Leisure time, View on life, Creativity, Learning, Friends and Friendship, and View of self) and provides a total score between 0 and 96 with a higher score representing a higher level of quality of life.
Negative effects | After the intervention.
  Negative effects of the treatment were assessed with a questionnaire comprising 12 items regarding common symptoms such as fatigue, dizziness, and negative mood
Sleep diary- Sleep onset latensy (SOL) | Baseline, daily through study completion, up to 8 weeks
  It is measured in minutes and calculated. The participant will register this in the sleep diary.
Sleep diary- wake after sleep onset (WASO) | Baseline, daily through study completion, up to 8 weeks
  It is measured in minutes and calculated. The participant will register this in the sleep diary.
Sleep diary. early morning awakening (EMA) | Baseline, daily through study completion, up to 8 weeks
  It is measured in minutes and calculated. The participant will register this in the sleep diary.
Multiple Sclerosis Impact Scale (MSIS-29) | Baseline (before the treatment) after the treatment that is 6 to 8 weeks after entering the treatment and 6 and 12 months after the treatment.
  The MSIS-29 measures physical and psychological impact of MS. Items on the MSIS-29 have a Likert scale format (range 1.00-5.00); higher scores indicate a greater degree of disability. Total score is derived by summing items and transforming them into a score out of 100; higher scores imply a greater degree of disability.
Client Satisfaction Questionnaire-8 (CSQ-8) | After the treatment that is 6 to 8 weeks after entering the treatment
  It is a brief global measure of client satisfaction..The CSQ-8 comprises eight items regarding service satisfaction that are scored on a 4-point Likert scale and provides a total score between 8 and 32. Higher values indicating higher satisfaction.

OTHER OUTCOMES:
The severity of MS - MS check | Screening
  The MS check which is a self-assessment questionnaire consisting of 14 questions concerning fatigue, cognition, mood, vision, speech/communication, and other bodily functions scored on a scale from 0 to 3. Higher scores indicating more severe disability and symptoms related to MS.
The Credibility/Expectancy Questionnaire | Will be administered after the first treament week.
  The questionnaire contains 6 items rated on a 1-9 or a 0%-100% scale, depending upon the item. In the credibility factor the items explore: if the treatment appears logical; if the treatment appears useful; and if the treatment is reliable.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Buhrman, phd, Principal Investigator — Uppsala University
Locations (1):
- Department of Psychology, Uppsala University, Uppsala, Uppland, Sweden